CLINICAL TRIAL: NCT02614547
Title: A Multicenter, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Study Evaluating The Efficacy, Safety, And Pharmacokinetics Of SAGE-547 Injection In The Treatment Of Adult Female Subjects With Severe Postpartum Depression
Brief Title: A Study to Evaluate SAGE-547 in Participants With Severe Postpartum Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 547-PPD-202 A
Record Dates: First submitted 2015-11-02; First posted 2015-11-25 (Estimated); Results first posted 2021-09-13 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2022-01

CONDITIONS: Severe Postpartum Depression
MeSH Terms: conditions — Depression, Postpartum | interventions — brexanolone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Participants received infusion rates of placebo matched to SAGE-547.
  Interventions: Drug: Placebo
- SAGE-547 (Experimental): Participants received a 4-hour dose titration of 30 micrograms per kilogram per hour (micrograms/kg/hr) (0 to 4 hours), then 60 micrograms/kg/hr (4 to 24 hours), then 90 micrograms/kg/hr (24 to 52 hours), followed by a taper to 60 micrograms/kg/hr (52 to 56 hours), and 30 micrograms/kg/hr (56 to 60 hours).
  Interventions: Drug: SAGE-547

INTERVENTIONS:
Drug: SAGE-547 — Administered as intravenous infusion.
  Arms: SAGE-547
Drug: Placebo — Administered as intravenous infusion.
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, parallel-group, placebo-controlled study of the efficacy, safety, and pharmacokinetics of SAGE-547 Injection in adult female participants diagnosed with severe postpartum depression.

ELIGIBILITY:
Key Inclusion Criteria:

* Participant either must have ceased lactating at Screening; or if still lactating at Screening, must have already fully and permanently weaned their infant(s) from breastmilk; or if still actively breastfeeding at Screening, must agree to cease giving breastmilk to their infant(s) prior to receiving study drug.
* Participant had a major depressive episode that began no earlier than the third trimester and no later than the first 4 weeks following delivery, as diagnosed by Structured Clinical Interview for DSM-IV Axis I Disorders (SCID-I).
* Participant was less than or equal to (<=) six months postpartum.
* Participant must be amenable to intravenous therapy.

Key Exclusion Criteria:

* Active psychosis.
* Attempted suicide associated with index case of postpartum depression.
* Medical history of seizures.
* Medical history of bipolar disorder.

Note: suicidal ideation was not an exclusion. Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2015-12-15 (Actual); Primary Completion 2016-06-22 (Actual); Study Completion 2016-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Kanes, MD, PhD, Study Chair — Sage Therapeutics
Locations (4):
- United States (4):
  - Sage Investigational Site, Atlanta, Georgia
  - Sage Investigational Site, Worcester, Massachusetts
  - Sage Investigational Site, Chapel Hill, North Carolina
  - Sage Investigational Site, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Data sharing will be consistent with the results submission policy of ClinicalTrials.gov.

REFERENCES:
- [Derived] Gerbasi ME, Meltzer-Brody S, Acaster S, Fridman M, Bonthapally V, Hodgkins P, Kanes SJ, Eldar-Lissai A. Brexanolone in Postpartum Depression: Post Hoc Analyses to Help Inform Clinical Decision-Making. J Womens Health (Larchmt). 2021 Mar;30(3):385-392. doi: 10.1089/jwh.2020.8483. Epub 2020 Nov 12. PMID 33181049
- [Derived] Kanes S, Colquhoun H, Gunduz-Bruce H, Raines S, Arnold R, Schacterle A, Doherty J, Epperson CN, Deligiannidis KM, Riesenberg R, Hoffmann E, Rubinow D, Jonas J, Paul S, Meltzer-Brody S. Brexanolone (SAGE-547 injection) in post-partum depression: a randomised controlled trial. Lancet. 2017 Jul 29;390(10093):480-489. doi: 10.1016/S0140-6736(17)31264-3. Epub 2017 Jun 12. PMID 28619476
- See also: Related Info — http://www.sagerx.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 4 centers in the United States from 15 December 2015 to 22 June 2016.
Pre-assignment Details: A total of 21 participants were randomized into the study to receive either placebo or SAGE-547.
Groups:
- SAGE-547: Participants received a 4-hour dose titration period of 30 micrograms per kilogram per hour (micrograms/kg/hr) (0 to 4 hours), then 60 micrograms/kg/hr (4 to 24 hours), then 90 micrograms/kg/hr (24 to 52 hours), followed by a taper to 60 micrograms/kg/hr (52 to 56 hours), and 30 micrograms/kg/hr (56 to 60 hours).
Period: Overall Study
Arm/Group | Placebo | SAGE-547
Started | 11 | 10
Completed | 11 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized population included the subset of participants from all enrolled population who were randomized.
Groups:
- SAGE-547: Participants received a 4-hour dose titration period of 30 micrograms/kg/hr (0 to 4 hours), then 60 micrograms/kg/hr (4 to 24 hours), then 90 micrograms/kg/hr (24 to 52 hours), followed by a taper to 60 micrograms/kg/hr (52 to 56 hours), and 30 micrograms/kg/hr (56 to 60 hours).
- Total: Total of all reporting groups
Arm/Group | Placebo | SAGE-547 | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.8 (4.58) | 27.4 (5.34) | 28.1 (4.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 7 | 13
  White | 5 | 3 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline at End of Treatment Period (at 60 Hours) in Hamilton Rating Scale for Depression (HAM-D) Total Score
Description: The HAM-D total score comprises a sum of the 17 individual item scores. Items scored in a range of 0 to 2 include: insomnia (early, middle, late), somatic symptoms (gastrointestinal and general), genital symptoms, loss of weight, and insight. The following items are scored in a range of 0 to 4: agitation, depressed mood, feelings of guilt, suicide, work and activities, retardation, anxiety (psychic and somatic), and hypochondriasis. The total score can range from 0 to 52, and higher scores indicate a greater degree of depression. A negative change from baseline indicates less depression. A positive change from baseline indicates more depression.
Time Frame: Baseline, 60 Hours
Population: Efficacy population included the subset of the all randomized participants who started the study drug infusion and who had a valid baseline HAM-D assessment and at least one post-baseline HAM-D assessment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | SAGE-547
Number analyzed (Participants) | 11 | 10
score on a scale | -8.75 (2.800) | -20.97 (2.938)
Statistical Analysis 1: Comparison: Placebo vs SAGE-547; Mixed Effects Model for Repeated Measure (MMRM) used an unstructured covariance model time points within participant. Fixed effects were treatment, baseline total score, assessment time point, and time point-by-treatment; Test type: Superiority; p = 0.008, MMRM; Least Squares Mean Difference = -12.22, 95% CI 2-sided [-20.77 to -3.67], Standard Error of Mean 4.081

2. Secondary Outcome: Percentage of Participants With HAM-D Response
Description: The HAM-D response was defined as having a 50 percent (%) or greater reduction from baseline in HAM-D total score. The HAM-D total score comprises a sum of the 17 individual item scores. Items scored in a range of 0 to 2 include: insomnia (early, middle, late), somatic symptoms (gastrointestinal and general), genital symptoms, loss of weight, and insight. The following items are scored in a range of 0 to 4: agitation, depressed mood, feelings of guilt, suicide, work and activities, retardation, anxiety (psychic and somatic), and hypochondriasis. The total score can range from 0 to 52, and higher scores indicate a greater degree of depression. A negative change from baseline indicates less depression. A positive change from baseline indicates more depression.
Time Frame: 60 Hours, Days 7 and 30
Population: Efficacy population included the subset of the all randomized participants who started the study drug infusion and who had a valid baseline HAM-D assessment and at least one post-baseline HAM-D assessment. Here, 'number analyzed' signifies participants evaluable for this outcome measure at specified time points.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | SAGE-547
Number analyzed (Participants) | 11 | 10
percentage of participants
  60 Hours | 36.4 | 70.0
  Day 7: number analyzed (Participants) | 10 | 10
  Day 7 | 20.0 | 80.0
  Day 30 | 27.3 | 70.0
Statistical Analysis 1: Comparison: Placebo vs SAGE-547; 60 Hours; Test type: Superiority; p = 0.198, Fisher Exact; Odds Ratio (OR) = 4.08, 95% CI 2-sided [0.49 to 37.67]
Statistical Analysis 2: Comparison: Placebo vs SAGE-547; Day 7; Test type: Superiority; p = 0.023, Fisher Exact; Odds Ratio (OR) = 16.00, 95% CI 2-sided [1.31 to 239.57]
Statistical Analysis 3: Comparison: Placebo vs SAGE-547; Day 30; Test type: Superiority; p = 0.086, Fisher Exact; Odds Ratio (OR) = 6.22, 95% CI 2-sided [0.70 to 62.08]

3. Secondary Outcome: Percentage of Participants With HAM-D Remission
Description: The HAM-D remission was defined as having a HAM-D total score of less than or equal to (<=)7. The HAM-D total score comprises a sum of the 17 individual item scores. Items scored in a range of 0 to 2 include: insomnia (early, middle, late), somatic symptoms (gastrointestinal and general), genital symptoms, loss of weight, and insight. The following items are scored in a range of 0 to 4: agitation, depressed mood, feelings of guilt, suicide, work and activities, retardation, anxiety (psychic and somatic), and hypochondriasis. The total score can range from 0 to 52, and higher scores indicate a greater degree of depression. A negative change from baseline indicates less depression. A positive change from baseline indicates more depression.
Time Frame: 60 Hours, Days 7, and 30
Population: Efficacy population included the subset of the all randomized participants who started the study drug infusion and who had a valid baseline HAM-D assessment and at least one post-baseline HAM-D assessment. Here, 'number analyzed'' signifies participants evaluable for this outcome measure at specified time points.
Measure: Number; unit: percentage of participants
Groups:
- SAGE-547: Participants received a 4-hour dose titration period of 30 (micrograms/kg/hr) (0 to 4 hours), then 60 micrograms/kg/hr (4 to 24 hours), then 90 micrograms/kg/hr (24 to 52 hours), followed by a taper to 60 micrograms/kg/hr (52 to 56 hours), and 30 micrograms/kg/hr (56 to 60 hours).
Arm/Group | Placebo | SAGE-547
Number analyzed (Participants) | 11 | 10
percentage of participants
  60 Hours | 9.1 | 70.0
  Day 7: number analyzed (Participants) | 10 | 10
  Day 7 | 0.0 | 70.0
  Day 30 | 18.2 | 70.0
Statistical Analysis 1: Comparison: Placebo vs SAGE-547; 60 Hours; Test type: Superiority; p = 0.008, Fisher Exact; Odds Ratio (OR) = 23.33, 95% CI 2-sided [1.56 to 1152.71]
Statistical Analysis 2: Comparison: Placebo vs SAGE-547; Day 7; Test type: Superiority; p = 0.003, Fisher Exact
Statistical Analysis 3: Comparison: Placebo vs SAGE-547; Day 30; Test type: Superiority; p = 0.030, Fisher Exact; Odds Ratio (OR) = 10.50, 95% CI 2-sided [1.01 to 140.57]

4. Secondary Outcome: Change From Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score
Description: The MADRS is a ten-item diagnostic questionnaire which psychiatrists use to measure the severity of depressive episodes in participants with mood disorders. It was designed as an adjunct to the HAM-D, to be more sensitive than the Hamilton Scale to the changes brought on by antidepressants and other forms of treatment. Each item yielded a score of 0 to 6. The MADRS total score was calculated as the sum of the 10 individual item scores, which ranged from 0 to 60. Higher MADRS scores indicate more severe depression. A negative change from baseline indicate less severe depression. A positive change from baseline indicates more severe depression.
Time Frame: Baseline, 60 Hours, Days 7 and 30
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | SAGE-547
Number analyzed (Participants) | 11 | 10
score on a scale
  Hour 60 | -12.10 (3.817) | -27.96 (4.001)
  Day 7: number analyzed (Participants) | 10 | 10
  Day 7 | -11.60 (3.766) | -27.56 (3.929)
  Day 30 | -11.19 (3.594) | -26.26 (3.767)
Statistical Analysis 1: Comparison: Placebo vs SAGE-547; 60 Hours: MMRM used an unstructured covariance model for time points within participant. Fixed effects were treatment, baseline total score, assessment time point, and time point-by-treatment; Test type: Superiority; p = 0.010, MMRM; Least Squares Mean Difference = -15.86, 95% CI 2-sided [-27.50 to -4.22], Standard Error of Mean 5.536
Statistical Analysis 2: Comparison: Placebo vs SAGE-547; Day 7: MMRM used an unstructured covariance model for time points within participant. Fixed effects were treatment, baseline total score, assessment time point, and time point-by-treatment; Test type: Superiority; p = 0.009, MMRM; Least Square Mean Difference = -15.96, 95% CI 2-sided [-27.43 to -4.50], Standard Error of Mean 5.448
Statistical Analysis 3: Comparison: Placebo vs SAGE-547; Day 30: MMRM used an unstructured covariance model for time points within participant. Fixed effects were treatment, baseline total score, assessment time point, and time point-by-treatment; Test type: Superiority; p = 0.010, MMRM; Least Square Mean Difference = -15.07, 95% CI 2-sided [-26.05 to -4.09], Standard Error of Mean 5.213

5. Secondary Outcome: Percentage of Participants With Clinical Global Impression-Improvement (CGI-I) Response
Description: The CGI-I item employs a 7-point Likert scale to measure the overall improvement in the participant's condition post-treatment. The investigator rated the participant's total improvement whether or not it was due entirely to drug treatment. Response choices include: 0 = not assessed, 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse. The CGI-I was only rated at post-treatment assessments, and by definition, was evaluated against baseline conditions. CGI-I response was defined as having a CGI-I score of "very much improved" or "much improved".
Time Frame: 60 Hours, Days 7 and 30
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Groups:
- Placebo: Participants received infusion rates of matching placebo identical to SAGE-547.
Arm/Group | Placebo | SAGE-547
Number analyzed (Participants) | 11 | 10
percentage of participants
  Hour 60 | 36.4 | 80.0
  Day 7: number analyzed (Participants) | 10 | 10
  Day 7 | 20.0 | 80.0
  Day 30 | 27.3 | 80.0
Statistical Analysis 1: Comparison: Placebo vs SAGE-547; 60 Hours; Test type: Superiority; p = 0.080, Fisher Exact; Odds Ratio (OR) = 7.00, 95% CI 2-sided [0.73 to 90.81]
Statistical Analysis 2: Comparison: Placebo vs SAGE-547; Day 7; Test type: Superiority; p = 0.023, Fisher Exact; Odds Ratio (OR) = 16.00, 95% CI 2-sided [1.31 to 239.57]
Statistical Analysis 3: Comparison: Placebo vs SAGE-547; Day 30; Test type: Superiority; p = 0.030, Fisher Exact; Odds Ratio (OR) = 10.67, 95% CI 2-sided [1.04 to 142.20]

6. Secondary Outcome: Change From Baseline in HAM-D Bech 6 Subscale
Description: The HAM-D Bech 6 subscale score was calculated as the sum of the following six items: depressed mood, feelings of guilt, work and activities, retardation, psychic anxiety, and general somatic symptoms. Each item is scored in a range of 0 to 2 or 0 to 4, with higher scores indicating a greater degree of depression. The scores were transformed to a scale of 0 to 100, with a higher score indicating a greater degree of depression. A negative change from baseline indicates less depression. A positive change from baseline indicates more depression.
Time Frame: Baseline, 60 Hours, Days 7 and 30
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | SAGE-547
Number analyzed (Participants) | 11 | 10
score on a scale
  60 Hours | -4.89 (1.701) | -10.94 (1.784)
  Day 7: number analyzed (Participants) | 10 | 10
  Day 7 | -3.99 (1.676) | -10.44 (1.754)
  Day 30 | -3.34 (1.772) | -10.14 (1.858)
Statistical Analysis 1: Comparison: Placebo vs SAGE-547; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.025, MMRM; Least Squares Mean Difference = -6.05, 95% CI 2-sided [-11.24 to -0.86], Standard Error of Mean 2.466
Statistical Analysis 2: Comparison: Placebo vs SAGE-547; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p = 0.016, MMRM; Least Squares Mean Difference = -6.46, 95% CI 2-sided [-11.57 to -1.34], Standard Error of Mean 2.427
Statistical Analysis 3: Comparison: Placebo vs SAGE-547; [analysis description as in outcome 4, analysis 3]; Test type: Superiority; p = 0.018, MMRM; Least Squares Mean Difference = -6.80, 95% CI 2-sided [-12.25 to -1.35], Standard Error of Mean 2.568

7. Secondary Outcome: Change From Baseline to 60 Hours in the HAM-D Individual Item Scores
Description: The HAM-D comprises individual ratings of the following symptoms scored in a range of 0 to 2: insomnia (early, middle, late), somatic symptoms (gastrointestinal and general), genital symptoms, loss of weight, and insight. The following symptoms are scored in a range of 0 to 4: agitation, depressed mood, feelings of guilt, suicide, work and activities, retardation, anxiety (psychic and somatic), and hypochondriasis. Higher scores indicate a greater degree of depression. A negative change from baseline indicates less depression. A positive change from baseline indicates more depression.
Time Frame: Baseline, 60 Hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | SAGE-547
Number analyzed (Participants) | 11 | 10
score on a scale
  Depressed Mood, Change From Baseline to 60 Hours | -1.4 (1.57) | -2.5 (1.58)
  Feeling of Guilt ,Change From Baseline to 60 Hours | -0.5 (0.69) | -1.7 (0.95)
  Suicide, Change From Baseline to 60 Hours | -0.4 (0.67) | -1.1 (0.88)
  Insomnia - Early, Change From Baseline to 60 Hours | -0.5 (0.69) | -1.6 (0.70)
  Insomnia -Middle, Change From Baseline to 60 Hours | -0.5 (0.69) | -1.6 (0.52)
  Insomnia - Late, Change From Baseline to 60 Hours | -0.4 (0.50) | -1.1 (0.74)
  Work and Activities, Change From Baseline to 60 Hours | -1.4 (1.36) | -2.4 (1.35)
  Retardation, Change From Baseline to 60 Hours | -0.5 (0.69) | -0.8 (0.79)
  Agitation, Change From Baseline to 60 Hours | -0.3 (0.65) | -0.3 (0.67)
  Anxiety-Psychic, Change From Baseline to 60 Hours | -0.9 (1.30) | -1.9 (1.29)
  Anxiety-Somatic, Change From Baseline to 60 Hours | -1.0 (1.10) | -1.9 (1.66)
  Gastrointestinal, Change From Baseline to 60 Hours | -0.4 (0.81) | -0.7 (0.95)
  Somatic General, Change From Baseline to 60 Hours | -0.4 (0.67) | -1.5 (0.85)
  Genital Symptoms, Change From Baseline to 60 Hours | -0.2 (0.60) | -0.8 (0.79)
  Hypochondriasis, Change From Baseline to 60 Hours | -0.3 (1.19) | -0.5 (0.71)
  Loss of Weight, Change From Baseline to 60 Hours | -0.4 (0.67) | -0.2 (0.67)
  Insight, Change From Baseline to 60 Hours | 0.0 (0.00) | 0.0 (0.00)

8. Secondary Outcome: Change From Baseline in Generalized Anxiety Disorder 7-item Scale (GAD-7) Total Score
Description: The GAD-7 is a participant-rated, generalized anxiety symptom severity scale. Scoring for GAD-7 generalized anxiety is calculated by assigning scores of 0 = "not at all sure," 1 = "several days," 2 = "over half the days," and 3 = "nearly every day" to the response categories. The GAD-7 total score for the seven items ranges from 0 to 21, where a score of 0 to 4 = minimal anxiety, 5 to 9 = mild anxiety, 10 to 14 = moderate anxiety, and 15 to 21 = severe anxiety. The GAD-7 total score was calculated as the sum of the seven individual item scores. A negative change from baseline indicates less anxiety. A positive change from baseline indicates more anxiety.
Time Frame: Baseline, 60 Hours, Day 7 and 30
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | SAGE-547
Number analyzed (Participants) | 11 | 10
score on a scale
  60 Hours | -9.08 (1.673) | -7.21 (1.757)
  Day 7: number analyzed (Participants) | 10 | 10
  Day 7 | -7.96 (1.986) | -9.44 (1.986)
  Day 30 | -7.38 (1.951) | -9.48 (2.050)
Statistical Analysis 1: Comparison: Placebo vs SAGE-547; 60 Hours; Test type: Superiority; p = 0.457, ANCOVA; Least Squares Mean Difference = 1.87, 95% CI 2-sided [-3.30 to 7.04], Standard Error of Mean 2.461
Statistical Analysis 2: Comparison: Placebo vs SAGE-547; Day 7; Test type: Superiority; p = 0.613, ANCOVA; Least Square Mean = -1.47, 95% CI 2-sided [-7.50 to 4.55], Standard Error of Mean -1.47
Statistical Analysis 3: Comparison: Placebo vs SAGE-547; Day 30; Test type: Superiority; p = 0.474, ANCOVA; Least Square Mean = -2.10, 95% CI 2-sided [-8.13 to 3.93], Standard Error of Mean 2.871

9. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it did not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A TEAE was defined as an AE with onset on or after the start of study drug infusion, or any worsening of a pre-existing medical condition/AE with onset on or after the start of study drug infusion.
Time Frame: Up to 30 days
Population: Safety population included all randomized participants who started the study drug infusion.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SAGE-547
Number analyzed (Participants) | 11 | 10
Participants | 8 | 4

ADVERSE EVENTS:
Time Frame: Up to 30 days
Description: Safety population included all randomized participants who started the study drug infusion.
Groups:
- SAGE-547: Participants received a 4-hour dose titration period of 30 microgram per kilogram per hour (microgram/kg/hr) (0 to 4 hours), then 60 microgram/kg/hr (4 to 24 hours), then 90 microgram/kg/hr (24 to 52 hours), followed by a taper to 60 microgram/kg/hr (52 to 56 hours), and 30 microgram/kg/hr (56 to 60 hours).
Arm/Group | Placebo | SAGE-547
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 8/11 | 4/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=11) | SAGE-547 (N=10)
Dizziness (Nervous system disorders) | 3 | 2
Somnolence (Nervous system disorders) | 0 | 2
Dizziness postural (Nervous system disorders) | 0 | 1
Sedation (Nervous system disorders) | 0 | 1
Abnormal dreams (Psychiatric disorders) | 2 | 0
Headache (Nervous system disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Tension headache (Nervous system disorders) | 1 | 0
Sinus Tachycardia (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Dry Mouth (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 1
Infusion Site Extravasation (General disorders) | 1 | 0
Infusion Site Pain (General disorders) | 2 | 0
Localised Odema (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Skin Abrasion (Injury, poisoning and procedural complications) | 1 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Hot Flush (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI can either be a party and subject to the same restrictions as the institution, or if not a party, the restrictions are described on the face of the contract (i.e., PI is a contractor of the institution; PI is part of a larger group of study personnel; institution has contracted with or otherwise bound all study personnel under confidentiality obligations and requirements to vest intellectual property to the institution).